CLINICAL TRIAL: NCT01473160
Title: DAILIES TOTAL1 Pre-Lens Tear Film Performance - Pilot Trial
Brief Title: Daily Disposable Contact Lens Tear Film Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Collaborators: Aston University (Other)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: P-347-C-014v2
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Results first posted 2013-01-16 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- delefilcon A (Experimental): Delefilcon A randomly assigned to one eye, with narafilcon A assigned to the fellow eye for contralateral wear. Both products will be worn for one day for 16 hours (+/- 1 hour).
  Interventions: Device: delefilcon A contact lens
- narafilcon A (Active Comparator): Narafilcon A randomly assigned to one eye, with delefilcon A assigned to the fellow eye for contralateral wear. Both products will be worn for one day for 16 hours (+/- 1 hour).
  Interventions: Device: narafilcon A contact lens

INTERVENTIONS:
Device: delefilcon A contact lens — CE-marked, silicone hydrogel, single vision, soft contact lens for daily disposable wear
  Other Names: DAILIES TOTAL1
  Arms: delefilcon A
Device: narafilcon A contact lens — Commercially marketed, silicone hydrogel, single vision, soft contact lens for daily disposable wear.
  Other Names: 1-DAY ACUVUE TruEye
  Arms: narafilcon A

SUMMARY:
The purpose of this study was to evaluate the pre-lens tear film stability of a new CE-marked daily disposable contact lens as compared to a commercially available daily disposable contact lens.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age of consent and sign Informed Consent document.
* Willing and able to wear spherical contact lenses for 16 hours.
* Willing and able to wear spherical contact lenses within the available range of powers.
* Best corrected spectacle visual acuity equal or better than 20/25 or 6/7.5.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Anterior segment infection, inflammation, or abnormality.
* Any use of systemic medications for which contact lens wear could be contraindicated.
* History of refractive surgery or irregular cornea.
* Currently enrolled in any clinical trial.
* Eye injury within twelve weeks prior to enrollment.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Aston University, Birmingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one study center in the UK.
Groups:
- Overall Study: All enrolled participants
Period: Overall Study
Arm/Group | Overall Study
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 31 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Corrected Visual Acuity of 0.0 or Better
Description: Corrected visual acuity was measured with a digitized logMAR (logarithm of the minimum angle of resolution) chart. A logMAR acuity of 0.0 is considered normal distance eyesight.
Time Frame: Up to 16 hours after lens insertion
Population: All enrolled participants
Measure: Number; unit: participants
Groups:
- Delefilcon A: Delefilcon A contact lens in one eye, with narafilcon A in the fellow eye, worn one day, 16 hours
- Narafilcon A: Narafilcon A contact lens in one eye, with delefilcon A in the fellow eye, worn one day, 16 hours
Arm/Group | Delefilcon A | Narafilcon A
Number analyzed (Participants) | 9 | 9
participants
  8 hours after lens insertion | 9 (0.079) | 9 (0.089)
  12 hours after lens insertion | 9 (0.058) | 9 (0.078)
  16 hours after lens insertion | 9 (0.079) | 9 (0.063)

2. Primary Outcome: Pre-Lens Noninvasive Tear Break-Up Time
Description: The pre-lens tear film is the layer of tears located on top of the contact lens (i.e., between the eye lid and the contact lens). The time required for a dry spot to appear on the corneal surface after blinking is referred to as the tear film break-up time. Circular images were projected onto the corneal surface using a CA-1000 topographer, and the tear film reflection was observed on a 30-inch flat panel monitor. PL-NITBUT was recorded at the first sign of image distortion. Three measurements were taken and averaged together. A higher number represents a lengthening in the tear film break up time.
Time Frame: Up to 16 hours after lens insertion
Population: All enrolled participants
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Delefilcon A | Narafilcon A
Number analyzed (Participants) | 9 | 9
seconds
  8 hours after lens insertion | 12.7 (5.3) | 11.3 (3.5)
  12 hours after lens insertion | 12.2 (5.9) | 13.8 (5.4)
  16 hours after lens insertion | 10.5 (4.5) | 10.1 (2.9)

3. Primary Outcome: Average Tear Meniscus Height
Description: The tear meniscus height, i.e., the distance between the line of reflection along the top of the tear prism to the edge of the eyelid, was measured by the investigator using a digital slit lamp.
Time Frame: Up to 16 hours after lens insertion
Population: All enrolled participants
Measure: Mean (Standard Deviation); unit: pixels
Arm/Group | Delefilcon A | Narafilcon A
Number analyzed (Participants) | 9 | 9
pixels
  8 hours after lens insertion | 28.0 (6.9) | 26.7 (8.2)
  12 hours after lens insertion | 26.0 (5.2) | 24.0 (7.7)
  16 hours after lens insertion | 28.7 (11.1) | 27.1 (10.8)

4. Primary Outcome: Average Ocular Surface Temperature
Description: Ocular surface temperature (OST) was recorded by the investigator using a dynamic, non-contact, infrared thermography camera. The average OST (encompassing the wear of a contact lens) was taken at the center of the cornea, at the temporal upper limbal area, and over the central 5 mm2 of the cornea, 2 seconds post-blink.
Time Frame: Up to 16 hours after lens insertion
Population: All enrolled participants
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Delefilcon A | Narafilcon A
Number analyzed (Participants) | 9 | 9
Degrees Celsius
  8 hours after lens insertion | 35.6 (0.8) | 35.3 (0.8)
  12 hours after lens insertion | 35.2 (0.8) | 35.2 (0.9)
  16 hours after lens insertion | 35.5 (0.8) | 35.3 (1.3)

5. Secondary Outcome: Subjective Comfort
Description: Overall comfort was assessed by the participant and recorded on a scale from 0 (poor) to 10 (excellent) in response to the question, "How comfortable is the lens feeling at present?"
Time Frame: Up to 16 hours after lens insertion
Population: All enrolled participants
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Narafilcon A
Number analyzed (Participants) | 9 | 9
Units on a scale
  8 hours after lens insertion | 9.1 (0.8) | 6.8 (2.3)
  12 hours after lens insertion | 9.0 (0.9) | 6.7 (2.1)
  16 hours after lens insertion | 9.1 (0.8) | 6.3 (2.5)

6. Secondary Outcome: Subjective Vision
Description: Overall vision was assessed by the participant on scale from 0 (poor) to 10 (excellent) in response to the question, "What is the quality of your vision with the lens at present?"
Time Frame: Up to 16 hours after lens insertion
Population: All enrolled participants
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Narafilcon A
Number analyzed (Participants) | 9 | 9
Units on a scale
  8 hours after lens insertion | 9.0 (1.3) | 7.8 (1.9)
  12 hours after lens insertion | 8.7 (1.4) | 7.8 (1.6)
  16 hours after lens insertion | 8.7 (1.3) | 8.0 (1.1)

7. Secondary Outcome: Number of Participants With Adequate Lens Fit
Description: Lens fit was assessed by the investigator with a biomicroscope (slit lamp).
Time Frame: Up to 16 hours after lens insertion
Population: All enrolled participants
Measure: Number; unit: Participants
Arm/Group | Delefilcon A | Narafilcon A
Number analyzed (Participants) | 9 | 9
Participants
  8 hours after lens insertion | 9 | 9
  12 hours after lens insertion | 9 | 9
  16 hours after lens insertion | 9 | 9

ADVERSE EVENTS:
Description: This reporting group includes all enrolled participants.
Arm/Group | Delefilcon A | Narafilcon A
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

LIMITATIONS AND CAVEATS:
Pilot study. Small number of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No